CLINICAL TRIAL: NCT06579248
Title: Study of a Novel Intraoral Hypothermia Device for Preserving Taste During Radiation Therapy for Squamous Cell Carcinoma of the Larynx
Brief Title: Intraoral Hypothermia Device for Preserving Taste During Radiation
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Farzan Siddiqui, Senior Staff Physician, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15529-01
Record Dates: First submitted 2024-07-23; First posted 2024-08-30 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Cancer; Taste Dysfunction; Radiation Therapy
MeSH Terms: conditions — Head and Neck Neoplasms; Taste Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraoral Hypothermia Device (Experimental): An intraoral hypothermia device will be used to cool the oral cavity while subject's receive radiation therapy.
  Interventions: Device: Intraoral Device

INTERVENTIONS:
Device: Intraoral Device — Device that circulates cooled water through the oral cavity.

SUMMARY:
Radiation therapy to the head and neck region is known to cause taste dysfunction. Preliminary studies showed that cooling normal structures may lower damage caused by radiation. The purpose of this research study is to see if it is feasible to use an intraoral cooling device during radiation treatments to preserve or lower the decline of taste function.

ELIGIBILITY:
Inclusion Criteria:

* Patients being treated with combination radiation therapy and chemotherapy (definitive) for locally advanced (AJCC 8th cT3-4 or cN+) squamous cell carcinoma of the larynx.
* Age ≥ 18.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Patients will engage in the informed consent process and provide study-specific informed consent prior to study entry and must be able to fill out toxicity and quality of life related questionnaires.
* Patients should be concurrently treated with any of the following chemotherapy drugs: cisplatin, carboplatin, and cetuximab.

Exclusion Criteria:

* Patients receiving other forms of therapy intended to reduce taste dysfunction.
* Patients with metastatic disease.
* Patient with allergies or hypersensitivity to materials in the intraoral bolus.
* Patients who have received prior chemotherapy or radiation therapy for head and neck cancer.
* Patients who decline to use or cannot tolerate the intraoral device.
* Patients who are current or recent (within 3 months of treatment initiation) cigarette smokers.
* Patients who are unable to complete the required forms; however, verbal completion is adequate if recorded on the form daily.
* Patients with uncontrolled serious illness including, but not limited to, ongoing or serious active infection requiring IV antibiotics for over 30 days, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia other than chronic, stable atrial fibrillation, immunocompromised state, significant hepatic insufficiency, significant hematological disease, and any serious or unstable psychological condition.
* Patients who are on any of the following medication that cannot find a suitable substitute during the study period: acetazolamide, maribavir (TAK-620, Phase 3 trial drug), eszopiclone, topiramate, captopril, lithium, procainamide, terbinafine, and amiodarone.
* Patients who have taste loss at baseline, assessed subjectively and objectively at the first encounter, will be excluded from the study and all analysis. They will be replaced with a new patient.
* Patients who have tested positive for COVID-19 during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in Dysgeusia | 6 months after RT completion
  Taste will be measured objectively using Burghart taste strips in five different concentrations of salty, sweet, sour, bitter, and umami. Taste will be assessed on a yes/no scale to reflect the ability to correctly identify taste category.
  Taste will be measured subjectively with a series of previously-validated, patient-reported taste-related questions. The questions comprise of a modified Chemotherapy-induced Taste Alteration Scale (CiTAS), one question from the Head and Neck Quality of Life questionnaire (HNQOL, question 2H) and one question from the University of Washington Head and Neck-specific Quality of Life questionnaire (UWQOL, question 9).
  The CiTAS uses a scale of 1-5, with 1 meaning taste is normal and 5 being unable to taste.
  The HNQOL uses a scale of 1-5, with 1 meaning taste is normal and 5 being unable to taste.
  The UWQOL uses a scale of 1-4, with 1 meaning taste is normal and 4 being unable to taste.
  Questionnaires are used together to quantify change in taste.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other researchers.